CLINICAL TRIAL: NCT06608823
Title: A Study to Assess Safety and Effectiveness of the JenaValve Trilogy™ Transcatheter Heart Valve System Versus Surgical Valve Replacement in Patients With Aortic Regurgitation
Brief Title: ARTIST: Aortic Regurgitation Trial Investigating Surgery Versus Trilogy™
Acronym: ARTIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JenaValve Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JVT24001
Record Dates: First submitted 2024-09-17; First posted 2024-09-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Aortic Regurgitation; Aortic Valve Insufficiency; Aortic Insufficiency
MeSH Terms: conditions — Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Transcatheter Aortic Valve Replacement (TAVR) (Experimental): Transcatheter Aortic Valve Replacement (TAVR) using the Trilogy THV System
  Interventions: Device: Transcatheter Aortic Valve Replacement (TAVR) using Trilogy THV System
- SAVR (Other): SAVR using commercially available surgical prosthetic valve
  Interventions: Device: SAVR

INTERVENTIONS:
Device: Transcatheter Aortic Valve Replacement (TAVR) using Trilogy THV System — Transcatheter Aortic Valve Replacement (TAVR) with Trilogy Device
  Arms: Transcatheter Aortic Valve Replacement (TAVR)
Device: SAVR — SAVR using commercially available surgical prosthetic valves.
  Arms: SAVR

SUMMARY:
To demonstrate non-inferiority of the Trilogy Transcatheter Heart Valve (THV) System compared with surgical aortic valve replacement (SAVR) for treatment of subjects with clinically significant native aortic regurgitation (AR)

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indication for AVR for native valve predominant AR defined as:

   1. Class I or II indication for AVR according to ACC/AHA or ESC/EACTS guidelines with moderate to severe or severe AR (Grade ≥3+) on transthoracic echocardiography, transesophageal echocardiography or cardiac MRI as assessed by the core laboratory OR
   2. AR severity that remains indeterminate despite core laboratory review of all imaging including at least one advanced imaging modality (TEE or cardiac MRI) AND evidence of left ventricular damage* from AR with unanimous agreement from the local heart team, an independent clinical evaluation committee and the CRB that the symptomatic subject (NYHA II or greater) will benefit from SAVR for AR
2. The subject is a candidate for TAVR using the Trilogy THV system and SAVR using a commercially approved bioprosthetic heart valve
3. Subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits
4. Subject meets the legal minimum age to provide informed consent based on local regulatory requirements

Exclusion Criteria:

1. Confirmed moderate (2+) or less AR severity by core laboratory evaluation
2. Estimated life expectancy of less than 24 months due to associated non- cardiac comorbid conditions
3. Subject is high-risk for SAVR as determined by the local heart team
4. Subject refuses SAVR as a treatment option
5. Subject refuses a blood transfusion
6. Subject is selected for aortic valve repair or aortic surgery
7. Marfan syndrome or other known connective tissue disease that would necessitate aortic root replacement/intervention
8. Subject unable to undergo pre-procedure CT scan analysis for annular sizing
9. Mitral or tricuspid disease, considered clinically significant, such that if randomized to surgery, repair or replacement would be expected.
10. Subject has a known hypersensitivity or contraindication to all anticoagulation/antiplatelet medications (or inability to be anticoagulated for the index procedure), nitinol, or sensitivity to contrast media which cannot be adequately pre-medicated
11. Hostile chest or conditions or complications from a prior surgery that would preclude safe reoperation (i.e., mediastinitis, radiation damage, chest wall abnormalities, adhesion of aorta or internal mammary artery (IMA) to the sternum)
12. Need for emergency surgery or TAVR for any reason
13. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or need for mechanical circulatory support
14. Ongoing sepsis or active infective endocarditis with ongoing antibiotic (including suppressive) therapy or positive blood cultures within 6 weeks
15. Cardiac resynchronization therapy (CRT) device implantation within 30 days of randomization
16. LVEF <25% according to core laboratory measurement of resting echocardiogram at time of screening
17. Moderate to severe or worse right ventricular dysfunction on resting echocardiogram according to core laboratory
18. Severe chronic liver disease (Child-Pugh C) or any active liver disease
19. Chronic Kidney Disease Stage 4 or 5 (<30 cc/min/1.73 m2 or dialysis)
20. Severe Pulmonary Hypertension (pulmonary arterial systolic pressure

    * amp;amp;gt;2/3 systemic systolic pressure)
21. Severe Chronic Obstructive Pulmonary Disease (COPD) with FEV1

    * amp;amp;lt;50% predicted or need for chronic supplementary oxygen
22. Blood dyscrasia as defined: leukopenia (WBC <3,000 Cells/μL), thrombocytopenia (platelet count <50,000 Cells/μL), or anemia (hemoglobin <9.0 g/dL) that is uncorrected prior to randomization
23. History of bleeding diathesis or coagulopathy that is not adequately treated
24. Active gastrointestinal bleeding precluding anticoagulation or antiplatelet therapy
25. Any condition considered a contraindication to mechanical circulatory support
26. Uncontrolled atrial fibrillation (i.e., resting heart rate >120 bpm)
27. Evidence of an acute myocardial infarction ≤30 days before the index AVR
28. Any percutaneous coronary or peripheral interventional procedure performed ≤30 days prior to AVR (Subjects with placement of coronary or peripheral stent(s) should be assessed for the ability to safely proceed with SAVR within the protocol timeframe)
29. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within six weeks of randomization
30. Prior stroke with residual modified Rankin Score ≥2
31. Stroke or transient ischemic attack (TIA) within 6 months of randomization
32. Body mass index (BMI) <20 or >50 kg/m2
33. Currently participating in a cardiovascular investigational drug or device trial and has not yet completed follow-up for the primary endpoint (excluding registries)
34. Severe cognitive decline (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits)
35. Other medical, social, or psychological conditions that in the opinion of the investigator preclude the subject from appropriate consent or adherence to the protocol required follow-up exams
36. Pregnancy or intent to become pregnant prior to completion of all protocol follow-up requirements
37. Anatomical exclusion criteria (ANY of the following):

    1. Congenital bicuspid, unicuspid or quadricuspid aortic valve verified by echocardiography or CCT core laboratory
    2. Native aortic annulus perimeter <66 mm or >90 mm per the core laboratory reading of baseline cardiac CT imaging
    3. Iliofemoral arteries with vessel characteristics unsuitable for sheath passage (e.g., calcification, tortuosity) as determined by the case review board (CRB)
    4. Significant abdominal or thoracic aortic disease (such as porcelain aorta, aneurysm, severe calcification, aortic coarctation) that would preclude safe passage of the delivery system or cannulation and aortotomy for SAVR
    5. According to the CRB, a combination of aortic root angulation (angle between the plane of the aortic valve annulus and horizontal plane/vertebrae), sinus size, and straight length of the aorta that will not allow safe device delivery and THV deployment
    6. Sinus of Valsalva anatomy that would prevent adequate coronary perfusion after valve implantation
38. According to core laboratory evaluation, severe aortic stenosis
39. Uncorrected hypertrophic obstructive cardiomyopathy
40. Echocardiographic or Multi-slice CT (MSCT) evidence of untreated intracardiac mass or vegetation
41. Left ventricular thrombus
42. Left atrial thrombus without continuous appropriate anticoagulation within 90 days of the study procedure
43. Complex coronary artery disease:

    1. Unprotected left main coronary artery disease ≥50%
    2. Syntax score >32 (in the absence of prior revascularization)
    3. Heart Team determines that optimal revascularization cannot be adequately performed with EITHER CABG at the time of SAVR OR PCI at least 30 days prior to THV implant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1016 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2036-02 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality | 12 months
  all-cause mortality at 12 months
All stroke | 12 months
  Number of patients that had stroke
unplanned cardiac rehospitalization | 12 months
  Number of patients who had unplanned cardiac rehospitalization

SECONDARY OUTCOMES:
Length of index hospitalization | pre-intervention/procedure surgery
  comparing TAVR length of index hospitalization with SAVR
Echocardiographic effective orifice area | 30 days
  comparing TAVR Echocardiographic effective orifice area with SAVR
Moderate or greater patient prosthesis mismatch as measured by echo | 30 days or immediately after the intervention/procedure
  comparing TAVR moderate or greater patient prosthesis mismatched with SAVR
Kansas City Cardiomyopathy Questionnaire Overall Summary (KCCQ-OS) | 30 days
  comparing change in KCCQ-OS in TAVR with SAVR. the minimum and maximum values vary based on the questionnaire. Higher scores mean better outcome.
Atrial fibrillation | 30 days
  comparing the onset atrial fibrillation in TAVR with SAVR
Cardiovascular rehospitalization | 30 days
  comparing the number of cardiovascular rehospitalizations in TAVR with SAVR
Composite primary endpoints | 30 days
  comparing the superiority of the composite primary endpoint and its components in TAVR with SAVR
Composite primary endpoints | 1 year
  comparing the superiority of the composite primary endpoint and its components in TAVR with SAVR
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 30 days
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 6 months
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 1 year
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 2 years
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 3 years
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 4 years
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 5 years
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 6 years
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 7 years
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 8 years
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 9 years
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 10 years
  Freedom of Major Adverse Cardiovascular and Cerebrovascular Events

CONTACTS AND LOCATIONS:
Overall Officials: Vinod H Thourani, MD, Principal Investigator — Piedmont Heart Institute; Torsten P Vahl, MD, Principal Investigator — Columbia University; Raj Makkar, MD, Principal Investigator — Cedars-Sinai Medical Center; Hendrik Treede, MD, Principal Investigator — Department of Cardiovascular Surgery Johannes-Gutenberg University
Locations (19):
- United States (19):
  - CPMC Sutter Health, Burlingame, California
  - Scripps Health, La Jolla, California
  - Cedar-Sinai Medical Center, Los Angeles, California
  - BayCare Health, Clearwater, Florida
  - HCA North Florida, Gainesville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Piedmont Healthcare, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Minneapolis Heart Institute Founcation, Minneapolis, Minnesota
  - Cumc/Nyph, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Ohio Health, Columbus, Ohio
  - Houston Methodist Research Institute, Houston, Texas
  - Baylor Scott & White Health, Plano, Texas
  - Intermountain Health, Murray, Utah
  - Intermountain Healthcare, Murray, Utah
  - Sentara Norfolk, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Chronic Severe Aortic Regurgitation: Should We Lower Operating Thresholds? — https://pubmed.ncbi.nlm.nih.gov/31545685/
- See also: Global longitudinal strain in chronic asymptomatic aortic regurgitation: systematic review — https://pubmed.ncbi.nlm.nih.gov/36472208/
- See also: 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines — https://pubmed.ncbi.nlm.nih.gov/33332150/